CLINICAL TRIAL: NCT04921878
Title: Safety, Tolerability, Pharmacokinetics and Efficacy of Mitoxantrone Hydrochloride Liposome Injection in Chinese Patients With Advanced Solid Tumors: A Multicenter, Open-label, Phase I Dose-escalation and Dose-expansion Study
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection in Chinese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-025
Record Dates: First submitted 2021-05-31; First posted 2021-06-10 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2021-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): Dose-escalation phase: Patients will receive mitoxantrone hydrochloride liposome injection followed by a 3-week DLT observation period. The initial dose of mitoxantrone hydrochloride liposome injection will be set as 24 mg/m2, and then the dose is sequentially escalated to 30 mg/m2, 36 mg/m2 and 40 mg/m2.
  Dose-expansion phase: After DLT observation, two to four dose cohorts will be selected for dose-expansion to further evaluate the safety and efficacy of mitoxantrone hydrochloride liposome injection.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome injection — Mitoxantrone hydrochloride liposome injection will be administered intravenously once every 3 weeks (a cycle) for a maximum of 6 cycles.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and efficacy of mitoxantrone hydrochloride liposome injection in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase I dose-escalation and dose-expansion study aimed to evaluate the safety, tolerability, pharmacokinetics and efficacy of mitoxantrone hydrochloride liposome injection. This study consists of two phases: dose-escalation phase and dose expansion phase. The dose-escalation phase will be conducted to determine the maximum tolerated dose (MTD) of mitoxantrone hydrochloride liposome injection in patients with advanced solid tumors based on a 3+3 design. Patients enrolled in this phase will receive mitoxantrone hydrochloride liposome injection followed by a 3-week DLT observation period. After DLT observation, two to four dose cohorts will be selected for dose-expansion to further explore the safety and efficacy of study drug according to the dose-escalation results. In the dose-expansion phase, patients will receive the study drug every 3 weeks (q3w, a cycle) until disease progression, intolerable toxicity, death, or withdrawal by investigator or patient decision (a maximum of 6 cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Patients fully understand and voluntarily participate in this study and sign informed consent;
2. Aged 18-65 years, without gender limitation;
3. Histologically or cytologically confirmed advanced solid tumors;
4. Patients with advanced solid tumors who have been judged by the investigator to be ineffective with conventional therapy or lacking effective treatment, including those for whom no current standard of care is available or for whom is unable to tolerate standard therapy, etc.;
5. At least one measurable lesion according to RECIST v1.1 at baseline;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
7. AEs from the previous treatment have resolved to ≤ Grade 1 based on CTCAE (except for the toxicity without safety risk judged by the investigator, such as alopecia, hyperpigmentation);
8. Adequate organ function defined as:

   * Absolute neutrophil count (ANC) ≥1.5*109/L (No G-CSF treatment within 2 weeks prior to the laboratory test);
   * Hemoglobin ≥ 90 g/L (No red blood cell transfusion within 2 weeks prior to the laboratory test);
   * Platelet count ≥ 100*109/L (No platelet transfusion within 2 weeks prior to the laboratory test);
   * Creatinine ≤1.5 upper limit of normal (ULN);
   * Total bilirubin ≤1.5 ULN;
   * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 3 ULN;
   * Coagulation: prothrombin time (PT) or International Normalization Ratio (INR) ≤1.5 ULN
9. Female patients must have a urine or blood HCG negative test before enrolment (except for menopause and hysterectomy); Patients and their partners must agree to use effective contraceptives measures during the study until 6 months after the end of the last dose.

Exclusion Criteria:

1. History of severe allergy to mitoxantrone hydrochloride or any excipients of the study drug;
2. Cerebral or meningeal metastases;
3. Life expectancy < 3 months;
4. Patients with chronic hepatitis B (HBsAg or HBcAb positive with HBV DNA ≥ 1000 IU/mL), chronic hepatitis C (HCV antibody positive with HCV RNA above the lower limit of detection of the study center), or human immunodeficiency virus (HIV) antibody positive;
5. Active bacterial, fungal or viral infections that require intravenous infusion treatment within 1 week prior to the first dose;
6. Any anticancer treatment within 4 weeks prior to the first dose (e.g., radiotherapy, targeted therapy, immunotherapy, endocrine therapy, etc.); Traditional Chinese medicine or proprietary Chinese medicine with an approved oncology indication within 2 weeks prior to the first dose;
7. Enrolled in any other clinical trials within 4 weeks prior to the first dose;
8. Patients underwent major surgery within 3 months prior to the first dose did not fully recover, or have a surgical schedule during the study period;
9. Serious thrombosis or thromboembolism as judged by the investigator within 6 months prior to screening;
10. History of additional malignant tumor within 3 years, except for locally curable cancer that has been cured, such as basal or squamous cell skin cancer or in situ prostate, cervical or breast cancer;
11. Patients with the following cardiac function defects:

    * Long QTc syndrome or QTc interval > 480 ms;
    * Complete left bundle branch block, II-III degree atrioventricular block;
    * Severe, uncontrolled arrhythmias requiring pharmacological treatment;
    * History of chronic congestive heart failure, NYHA ≥ grade 3;
    * Cardiac ejection fraction < 50% within 6 months prior to screening;
    * Heart valve disease with CTCAE ≥ grade 3;
    * Uncontrollable hypertension (defined as a measured systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg under pharmacological control);
    * ECG evidence of myocardial infarction, unstable angina, history of severe pericardial disease, and acute ischemic or severe conduction system abnormalities within 6 months prior to screening;
12. Previous treatment with adriamycin or other anthracyclines, with the total cumulative dose (doxorubicin equivalent) >350 mg/m2;
13. Lactating female;
14. Serious and/or uncontrolled medical condition that, in the judgment of the investigator, may affect the patient's participation in this study (including, but not limited to: diabetes not effectively controlled, kidney disease requiring dialysis, severe liver disease, life-threatening autoimmune and bleeding disorders, substance abuse, neurological disorders, etc.);
15. Not suitable for this study as decided by the investigator due to other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Dose Limit toxicity (DLT) | Up to 21 days after the first dose
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From the initiation of the first dose to 28 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetic profile: Cmax | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Peak Plasma Concentration (Cmax)
Pharmacokinetic profile: Tmax | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Time to reach maximum concentration (Tmax)
Pharmacokinetic profile: AUC0-t | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUC0-t)
Pharmacokinetic profile: AUC0-∞ | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-∞)
Pharmacokinetic profile: t1/2 | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Half-time (t1/2)
Pharmacokinetic profile: CL | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Clearance (CL)
Pharmacokinetic profile: Vz | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Volume of Distribution (Vz)
Objective response rate (ORR) | Through study completion, an average of 2 years
  ORR is defined as the proportion of patients who have a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
Disease control rate (DCR) | Through study completion, an average of 2 years
  DCR is defined as the proportion of patients who have a response of CR/PR or stable disease (SD) as per RECIST 1.1
Duration of response (DoR) | Through study completion, an average of 2 years
  DoR is defined as the time from the first assessment of CR or PR until the date of first occurrence of progressive disease (PD) as per RECIST 1.1 or death from any cause, whichever occurs first
Progression-free survival (PFS) | Through study completion, an average of 2 years
  PFS is defined as the time from the date of first dose until the date of first documented PD as per RECIST 1.1 or death from any cause, whichever occurs first
Overall survival (OS) | Through study completion, an average of 2 years
  OS is defined as the time from the date of first dose until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Aimin Zang, Master, Principal Investigator — Affiliated Hospital of Hebei University
Locations (1):
- Affiliated Hospital of Hebei University, Baoding, Hebei, China